CLINICAL TRIAL: NCT00756145
Title: The Use of Low Molecular Weight Heparin in Hemodiafiltration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2008/421
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Kidney Disease
Keywords: stage V; treated; hemodiafiltration
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Injection of LMWH at the start of the hemodiafiltration session, at the inlet bloodline
  Interventions: Procedure: At start of the session, at the inlet line
- 2 (Experimental): Injection of LMWH 5 minutes after the start of the hemodiafiltration session, at the inlet bloodline
  Interventions: Procedure: 5 minutes after the start of the session, at the inlet line
- 3 (Experimental): Injection of LMWH at the start of the hemodiafiltration session, at the outline bloodline
  Interventions: Procedure: At the start of the session, at the outlet line

INTERVENTIONS:
Procedure: At start of the session, at the inlet line — Injection of LMWH at the inlet line, at the start of the hemodiafiltration session
  Arms: 1
Procedure: 5 minutes after the start of the session, at the inlet line — Injection of LMWH at the inlet line, 5 minutes after the start of the hemodiafiltration session
  Arms: 2
Procedure: At the start of the session, at the outlet line — Injection of LMWH at the outlet line, at the start of the hemodiafiltration session
  Arms: 3

SUMMARY:
Low molecular weight heparin (LMWH) is injected in the dialysis circuit at the start of the session. In the present study we compare 3 different methods of injection of LMWH: parameters of dialysis efficiency and clotting are measured. The study lasts 3 sessions for each patient.

ELIGIBILITY:
Inclusion Criteria:

* chronic kidney disease stade V treated with hemodiafiltration
* age >18 year
* Hematocrit > 30%

Exclusion Criteria:

* treatment with vitamin K antagonists
* treatment with other anti-coagulants or heparin besides the heparin used during dialysis
* active bleeding, infection or malignancy
* heparin associated allergy
* hepatic failure
* trombocytopenia < 120.000/µl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Anti-Xa activity at the end of the session | 240 min after start

SECONDARY OUTCOMES:
Anti-Xa activity during the session | at start, 30 min, 120 min and 180 min
ETP during the session | at start, 30 min, 120 min, 180 min and 240 min
Reduction ratio of urea | after 10min, 180min and 240min
Reduction ratio of beta2microglobulin | after 10min, 180min and 240min
Visual inspection of membrane and circuit | After the hemodiafiltration session
pressure measurements along the circuit | during the session
  inlet blood line, prefilter, transmembrane, outlet blood line

CONTACTS AND LOCATIONS:
Overall Officials: Annemieke Dhondt, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593
- [Derived] Dhondt A, Pauwels R, Devreese K, Eloot S, Glorieux G, Vanholder R. Where and When To Inject Low Molecular Weight Heparin in Hemodiafiltration? A Cross Over Randomised Trial. PLoS One. 2015 Jun 15;10(6):e0128634. doi: 10.1371/journal.pone.0128634. eCollection 2015. PMID 26076014
- See also: Website of the University Hospital Ghent — http://www.uzgent.be